CLINICAL TRIAL: NCT02289287
Title: Effects of a Self-Management Group-Intervention on Participation in Post-Stroke Patients.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulties in recruitment and academic time constrains we terminated the study after 60 participants instead of 90 as planned.
Sponsor: Uzi Milman (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Sponsor-Investigator, Uzi Milman, Director, Clinical Research Unit, Clalit Health Services, Haifa and Western Galilee District and the Department of Family Medicine, Faculty of Medicine, Technion- Israel Institute of Technology, HAIFA, ISRAEL, Clalit Health Services
Organization: Clalit Health Services (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COM - 0018-14-CTIL
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Stroke
Keywords: Self-Management; Stroke; Intervention; Group Processes
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Management group-intervention (Experimental): Participants will receive Self-Management group-intervention + Standard Care
  Interventions: Behavioral: Self-Management group-intervention
- Standard Care (Active Comparator): Participants will receive Standard Care only
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Self-Management group-intervention — At enrollment eligible patients will be randomized to Intervention + Standard Care or Standard Care group. Within 3 weeks after enrollment all participants will undergo baseline assessment using a predefined set of scales and questionnaires (intervention group will additionally undergo a semi-structured interview). The group-intervention (SM program) will begin after enrollment of at least 4 participants to the intervention group, and within no longer than 5 weeks since enrollment. The intervention will include 12 weekly sessions, each session 2.5 hour long, and will be based on well-known SM interventions that were found effective for stroke patients in the U.S. Follow-up assessments will be done at 12 and 36 week to examine long term effectiveness.
  Arms: Self-Management group-intervention
Behavioral: Standard Care — At enrollment eligible patients will be randomized to Intervention + Standard Care or Standard Care group. Within 3 weeks after enrollment all participants will undergo baseline assessment using a predefined set of scales and questionnaires (intervention group will additionally undergo a semi-structured interview). Standard care will include 'one-on-one' sessions in each paramedical discipline as given regularly in this setting (average of 15-20 sessions per patient). Follow-up assessments will be done at 12 and 36 week to examine long term effectiveness.
  Arms: Standard Care

SUMMARY:
Stroke is defined as a sudden vascular accident that causes brain damage and neurological impairment. Literature shows that a stroke has a negative effect on participation. Self-Management (SM) is defined as health promotion and education programs used mostly for people with chronic diseases, which aim at helping patients to maintain a feeling of wellness. The primary aim of this study is to assess the effectiveness of a group-based SM program for post-stroke patients in a community setting, and its contribution to improving participation, compared to standard care.

DETAILED DESCRIPTION:
At enrollment eligible patients will be randomized to Intervention + Standard Care or Standard Care group. Within 3 weeks after enrollment all participants will undergo baseline assessment using a predefined set of scales and questionnaires (intervention group will additionally undergo a semi-structured interview). The group-intervention (SM program) will begin after enrollment of at least 4 participants to the intervention group, and within no longer than 5 weeks since enrollment. The intervention will include 12 weekly sessions, each session 2.5 hour long, and will be based on well-known SM interventions that were found effective for stroke patients in the U.S. Standard care will include 'one-on-one' sessions in each paramedical discipline as given regularly in this setting (average of 15-20 sessions per patient). Follow-up measures will be performed within a week after the end of the intervention, and 6 months thereafter, in order to examine long term effectiveness. Outcome measures are questionnaires; change will be assessed by the difference in total score between T1 |(pre-intervention), T2 (post-intervention) and T3 (after 6 months)

ELIGIBILITY:
Inclusion Criteria:

Cerebrovascular accident diagnosed 3-18 months before enrollment. Treated at th Neurologic Rehabilitation Center of Clalit Health Services in Kiryat Byalik, Israel.

Living in the community (in their homes). Are capable of basic communication in Hebrew.

Exclusion Criteria:

Moderate-severe stroke (National Institutes of Health Stroke Scale (NIHSS) score ≤ 16).

Moderate-Severe Cognitive impairment (Montreal Cognitive Assessment (MOCA) - total score ≤ 16). Inability to provide informed consent.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Patient Participation | 12 and 36 weeks
  The primary outcome measure is the change in patient's participation, as defined by the International Classification of Function, Disability and Health (ICF), between the three assessment points - baseline, 12 and 36 weeks.

SECONDARY OUTCOMES:
Self-efficacy for self-management behaviors. | 12 and 36 weeks
  Self-efficacy for self-management behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Adar, MD, Principal Investigator — Clinical Research Unit, Clalit Health Services, Haifa District, HAIFA, ISRAEL; Eli Carmeli, PhD, Study Chair — Department of Physical Therapy, Faculty of Social Well fare and Health Sciences, Haifa University, Haifa, Israel.; Hagit Harel-Katz, MSc, Principal Investigator — Clinical Research Unit, Clalit Health Services, Haifa District, HAIFA, ISRAEL; Uzi Milman, MD, Study Director — Clinical Research Unit, Clalit Health Services, Haifa District, HAIFA, ISRAEL
Locations (1):
- Clinical Research Unit, Clalit Health Services, Haifa and Western Galilee District,, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harel-Katz H, Adar T, Milman U, Carmeli E. Examining the feasibility and effectiveness of a culturally adapted participation-focused stroke self-management program in a day-rehabilitation setting: A randomized pilot study. Top Stroke Rehabil. 2020 Dec;27(8):577-589. doi: 10.1080/10749357.2020.1738676. Epub 2020 Mar 14. PMID 32174261